CLINICAL TRIAL: NCT04978532
Title: The Effect of Guided Imagery Method on Procedural Pain in Children: A Randomized Controlled Trial
Brief Title: Effect of Guided Imagery Method on Procedural Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assistant Professor, PhD, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2021-07-03; First posted 2021-07-27 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Procedural Pain; Pain, Acute
Keywords: guided imagery; pain management; procedural pain; venipuncture
MeSH Terms: conditions — Pain, Procedural; Acute Pain; Agnosia | interventions — Imagery, Psychotherapy; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery Group (Experimental): One minute before venipuncture and during venipuncture, the children in the guided imagery group listened to a voice recording prepared in a studio. This voice recording named 'Stroll in the Forest' helped the children to imagine that they are strolling in a forest and guided them.
  Interventions: Other: Guided Imagery
- Control Group (Other): No intervention was performed to reduce pain in the control group.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Guided Imagery — The children in the guided imagery group listened to a voice recording named 'Stroll in the Forest' before and during venipuncture. One minute before venipuncture, children wore an earphone and voice recording started. Children closed their eyes, imagined the text content, and focused on the voice recording while listening to the voice. It is a voice recording that helps the children in the guided imagery group to imagine that they are strolling in a forest and guides them.
  Arms: Guided Imagery Group
Other: Control Group — No intervention was made in the children.
  Arms: Control Group

SUMMARY:
The study was conducted as a randomized controlled experimental trial. The children who attended a pediatric surgical clinic for venipuncture divided into two groups via randomization in the computer environment. After the randomization, the children in the guided imagery group listened to a voice recording prepared in a studio during venipuncture. This voice recording named 'Stroll in the Forest' helped the children to imagine that they are strolling in a forest and guided them. On the other hand, no application was performed on the children in the control group during the venipuncture. The primary outcome of the study was pain and secondary outcomes were heart rate and oxygen saturation values. The pain was evaluated by the children, parents, and observer. The pulse and oxygen saturation values were measured before, during, and after the venipuncture.

DETAILED DESCRIPTION:
Various nonpharmacological methods are used in reducing the pain of children. One of these non-pharmacological methods is the guided imagery method. In the guided imagery method, the imagination of children is used. It is possible to have children imagine by being guided with audible stimulus and, therefore, distract their attention from the procedure or pain/discomfort feeling. The aim of this study was to determine the effect of the guided imagery method on procedural pain level, heart rate, and oxygen saturation values of the children within the age range of 8-12 years. The sample size of the study has been determined by the power analysis (G*Power 3.1.9.2), in line with the results obtained from the studies which have been conducted using a similar research method. The sample size was found to be a total of 144 children including minimum of 72 children for each group. It was estimated that case losses may occur and therefore, it was decided to conduct the study with a total of 154 children including 77 children in two groups. One child in the guided imagery group was excluded from the study as he/she gave up listening to voice recording during the procedure and 1 child whose procedure could not be completed at once. In the control group, 1 child who felt nauseous during the procedure and 1 child whose procedure could not be completed at once could not be included in the sample group. Therefore, the sample group was composed of a total of 150 children including 75 children in each group. Information Form, Faces Pain Scale-Revised (FPS-R), and Visual Analogue Scale (VAS) were used for data collection.

Children and their parents who applied to the clinic for venipuncture were informed about the study. information about children and their parents included in the study were asked by the researcher through face-to-face interview and these data were recorded in 'Information Form' ten minutes before the procedure. FPS-R was explained to the children and they were asked whether or not they had pain before the procedure and they were asked to perform marking on the scale. Also, the children were told that they would mark the pain score again after the procedure. The parent was informed about 10-point VAS. Parent and observer (healthcare professional) marked children's pain level on the VAS independently by using a ruler. The researcher measured and recorded the pain level on the information form. The pulse oximeter device was attached to the finger of the extremity of the child that was not used for blood drawing. The children in the guided imagery group were informed that they would start to listen to voice recording named 'Stroll in the Forest' before venipuncture and blood would be drawn while they were listening to the voice recording. Also, children were asked to close their eyes, imagine the text content, and focus on the voice recording while listening to the voice. Thus, it was aimed to distract the children's attention from the procedure. One minute before venipuncture, children wore an earphone and voice recording started. As routine venipuncture procedure would be performed for the children in the control group, they were informed about the venipuncture procedure. Pre-procedure heart rate and oxygen saturation values of the children in the guided imagery group were determined and recorded just before attachment of tourniquet at the 50th second of the voice recording and then tourniquet was attached and blood drawing was started. Heart rate and oxygen saturation values of the children in the control group before attaching the tourniquet were written and then tourniquet was attached and then venipuncture was conducted. The blood of all the children included in the study was drawn by the experienced laboratorian working in the clinic using the 21 G needle-type injector. There was needle insertion in both control and guided imagery groups and when the first blood was seen in injector, the heart rate and oxygen saturation were recorded. Immediately after the injector was removed, the heart rate and oxygen saturation were recorded. Just after the procedure, children were asked to mark the pain level they felt during the procedure on FPS-R. The parent and observer evaluated the pain level of the children during the procedure using VAS.

ELIGIBILITY:
Inclusion Criteria:

* Speaking Turkish as a native speaker by children and parents,
* Being between the ages of 8 and 12,
* Not taking an analgesic, antipyretic, and anti-inflammatory drug within last 6 hours,
* Having body temperature at normal level (36.5-37.2⁰C),
* Having no disease that can cause chronic pain,
* Having no auditory, mental, and neurological disability that can affect their participation,
* Having no negative symptom-history during previous venipuncture,
* Having no allergy to strawberry included in the guided imagine text, and having no fear about forests and squirrels.

Exclusion Criteria:

* Not speaking Turkish as a native speaker by children and parents,
* Being younger than 8 years old and older than 12 years old,
* Taking an analgesic, antipyretic, and anti-inflammatory drug within last 6 hours,
* Having body temperature at a higher than normal level,
* Having a disease that can cause chronic pain,
* Having auditory, mental, and neurological disability that can affect their participation,
* Having negative symptom-history during previous venipuncture,
* Having allergy to strawberry included in the guided imagine text, and having fear about forests and squirrels.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Change of pain from before venipuncture to after venipuncture (assessed by children) | Before venipuncture procedure and after venipuncture procedure (immediately after the injector was removed)
  Pain assessed by children with Faces Pain Scale-Revised (FPS-R). This self-report scale is used to determine the level of acute pain. This scale is suitable for the use of children in the age range of 4-16 years and it is a commonly preferred valid and reliable scale. The scale is composed of a total of 6 facial expressions, rated from 0 to 10, starting from a neutral face expression (0 point) and including a picture of a face expressing the existence of severe pain without tears (10 points).
Change of pain from before venipuncture to after venipuncture (assessed by parents and the observer) | Before venipuncture procedure and after venipuncture procedure (immediately after the injector was removed)
  Pain assessed by parents and the observer with Visual Analog Scale (VAS). VAS is composed of a 100-mm horizontal line and the point "0" of this line expresses "no pain" and the point "10" expresses "worst pain". Firstly, the individual marks the intensity of the pain he/she perceives and the point marked by him/her is measured by using a ruler so that the pain score is determined

SECONDARY OUTCOMES:
Heart Rate | Before venipuncture procedure, during venipuncture procedure (when needle insertion and the first blood was seen in injector, until needle removed), and after venipuncture procedure (immediately after the injector was removed)
  Fingertip 'Creative' pulse oximeter device calibrated to measure the heart rate value of the children was used.The heart rate of all the children in the guided imagery group and control group recorded before, during, and after the venipuncture procedure.
Oxygen Saturation | Before venipuncture procedure, during venipuncture procedure (when needle insertion and the first blood was seen in injector, until needle removed), and after venipuncture procedure (immediately after the injector was removed)
  Fingertip 'Creative' pulse oximeter device calibrated to measure the oxygen saturation value of the children was used.The oxygen saturation of all the children in the guided imagery group and control group recorded before, during, and after the venipuncture procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Erkut, PhD, Principal Investigator — Biruni University; Duygu Gözen, PhD, Principal Investigator — Istanbul University Cerrahpaşa Florence Nightingale Faculty of Nursing
Locations (1):
- İstanbul University, Istanbul, Turkey (Türkiye)